CLINICAL TRIAL: NCT04006977
Title: Multistrain Probiotic Product (De Simone Formulation) Reduces Depression and Anxiety Scores: a Randomized Pilot Study in Patients With Ulcerative Colitis
Brief Title: Multistrain Probiotics Reduces UC Depression and Anxiety Scores
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Collaborators: MENDES SA (Unknown)
Responsible Party: Principal Investigator, Jie Liang, Professor of Gastroenterology Dept., Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XijingHDD-UC-Probiotics
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Ulcerative Colitis
Keywords: probiotics; psychological disorder;DSF
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: placebo plus standard therapy (Placebo Comparator): placebo plus standard therapy
  Interventions: Dietary Supplement: Placebo
- Arm 2: DSF plus standard therapy (Experimental): DSF (4 sachets/day) plus standard therapy
  Interventions: Dietary Supplement: a multistrain probiotic product (DSF)

INTERVENTIONS:
Dietary Supplement: a multistrain probiotic product (DSF) — In Arm 2, participants will receive standard medical therapy plus the multistrain probiotics (DSF), 4 sachets per day.
  Other Names: De Simone Fomulation (DSF), previously known as VSL#3 and now available as Vivomixx in EU and Visbiome in USA
  Arms: Arm 2: DSF plus standard therapy
Dietary Supplement: Placebo — In Arm 1, participants will receive standard medical therapy plus the placebo.
  Arms: Arm 1: placebo plus standard therapy

SUMMARY:
This pilot study aims to evaluate the effect of a 16-week duration of multistrain probiotic product (De Simone Fomulation (DSF), previously known as VSL#3 and now available as Vivomixx in EU and Visbiome in USA to reduce anxiety and depression scores in mild to moderate active UC. It has been known that gut microbiota is associated with IBD and mental health. In addition, IBD patients complicated with psychiatric disorders are rising more and more attention. Further, a recent study "Probiotic Bifidobacterium longum NCC3001 Reduces Depression Scores and Alters Brain Activity: A Pilot Study in Patients With Irritable Bowel Syndrome" was published in Gastroenterology in 2017, thus we wonder if DSF have an effect on the depression/anxiety in patients with UC）A total of 60 patients will be randomly allocated into two groups, group A will receive standard medical therapy plus placebo (4 sachets/day,), and group B will receive standard medical therapy plus DSF (each sachet containing 450 billion CFU, eight bacterial strains 4 sachets/day) for 16 weeks. The primary endpoint is the reduction of anxiety and depression scores after treatment (at 8 weeks and 16 weeks) using hospital anxiety and depression scale (HADS). The secondary endpoints including clinical response after 8-week and 16-week treatment (measured by a ≥3-point reduction in a Simple Clinical Colitis Activity Index (SCCAI) score at 16 weeks), and clinical remission (defined as SCCAI score ≤5 at 8 weeks and 16 weeks). Changes in fecal-associated microbiota by 16S ribosomal RNA sequencing and metabolomics using company service following probiotics therapy (at 16 weeks) were also assessed, stratified by both change in SCCAI score following probiotics therapy and randomization. Adverse events were evaluated at week 8 and 16 weeks by patient survey

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18
2. Patients with mild-to-moderately active UC (defined as a SCCAI score of ≥ 5 and < 12 and a colonoscopy will be performed to confirm the classification)
3. Patients with psychological dysfunction at screening based on hospital anxiety and depression scale (HADS), defined as HAD-A or HAD-D score ≥ 8
4. Signed Informed Consent obtained

Exclusion Criteria:

1. Severe ulcerative colitis (SCCAI score ≥ 12) or toxic dilatation of the colon
2. Prior bowel (either intestine or colon) resection surgery
3. Patients with any other disease or condition which might interfere with their participation in the trial, including significant hepatic, renal, endocrine, respiratory, neurologic, immune deficiency, cardiovascular, malignant diseases, bleeding disorders, autoimmune diseases and schizophrenia.
4. Take the following treatment:

   1. Antibiotics within 4 weeks prior to screening
   2. Oral steroids within the past 4 weeks before screening
   3. Acetyl-salicylic acid ≤100 mg/day as anti-platelet therapy or NSAIDs within 4 weeks prior screening
   4. Consecutive consumption of probiotics in 4 weeks prior to enrollment
   5. Topical or oral steroids within the past 4 weeks before screening
5. Patients requiring hospitalization or imminent need for surgery
6. Significant hepatic function abnormalities, defined as the values of serum ALT or AST ≥twice of the upper limit of normal value
7. Women who are planning or actual pregnancy or lactating during study period
8. Alcohol addiction (>40 g of alcohol/day，equivalent to >1 L of beer/day, 0.5 L of wine/day)
9. Patients with a history of a psychiatric condition other than anxiety or depression, use of opioids, antidepressants or anxiolytics in regular doses, illicit drug consumption
10. Patients participating or having participated in another clinical study 30 days prior to screening
11. Patients with one or more of the diseases: bacillary dysentery, amebic dysentery, chronic schistosomiasis, intestinal tuberculosis and Crohn's disease
12. Patients who are unwilling to comply with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
reduction of anxiety and depression scores | 0 week, 8 weeks, 12 weeks, 16 weeks
  reduction of anxiety and depression scores (with points as standard units) using HADS at 8 weeks and 16 weeks after randomized treatment

SECONDARY OUTCOMES:
Clinical response | 4 weeks, 8 weeks, 12 weeks, 16 weeks
  measured by a ≥1.5(3) points reduction in Simple Clinical Colitis Activity Index score at week 8 and 16
Clinical remission | 4 weeks, 8 weeks, 12 weeks, 16 weeks
  measured by Simple Clinical Colitis Activity Index score ≤5(2) points at week 8 and 16
Endoscopic remission/response | 0 week, 16 weeks
  measured by a Mayo endoscopic subscore of <1 point, or at least a 1 point reduction from baseline in the endoscopy subscore at week 16
Changes in fecal-associated microbiota following probiotic therapy | 0 week, 16 weeks
  Changes in fecal-associated microbiota using16S ribosomal RNA sequencing and changes in the metabolomic profile of the feces following probiotic therapy (at baseline and 16 weeks) will be assessed, stratified by both change in Simple Clinical Colitis Activity Index score following probiotic therapy and randomization.
Identification of potential stressors | 0 weeks, 16 weeks
  Participants will be asked to complete a modified practical and family problem list to identify 13 potential stressors.
Adverse events | 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Adverse events were assessed at week 8 and 16 by patient survey.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Liang, Professor, Principal Investigator — Hospital of Digeetive Disease, Xi'an, Shaanxi, Xijing, China
Locations (1):
- Xijing Digestive Disease, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Liu X, Zhou H, Zhang J, Li R, Liang J. Brain-gut co-management: probiotic LAB improves mental health and further reduces disease activity in ulcerative colitis patients with emotional disturbance. Nutr Neurosci. 2025 Dec;28(12):1511-1522. doi: 10.1080/1028415X.2025.2527224. Epub 2025 Jul 9. PMID 40629893